CLINICAL TRIAL: NCT06430229
Title: Evaluation of Atelectasis Frequency in Different Ventilation Modes Used in General Anesthesia in Children With Lung Ultrasonography
Brief Title: Atelectasis Frequency in Different Ventilation Modes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Aras, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AEŞH-BADEK-2024-152
Record Dates: First submitted 2024-05-09; First posted 2024-05-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Atelectasis; Mechanical Ventilation Complication; General Anesthesia; Lung Ultrasound
Keywords: Pulmonary Atelectasis; Mechanic Ventilation; General anesthesia; Lung Ultrasound
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients ventilated with volume controlled ventilation (VCV) mode (Active Comparator): Patients to be ventilated with VCV mode were placed on respiratory support (Dräger Primus) with a breathing rate that would provide 8 ml/kg tidal volume, 5 cmH2O positive end expiratory pressure (PEEP), and 30-35 mmHg end-tidal carbon dioxide concentration (etCO2) level.
  Interventions: Procedure: Volume controlled ventilation (VCV) mode
- Patients ventilated with pressure controlled ventilation (PCV) mode (Active Comparator): Appropriate peak inspiratory pressure was set to create a tidal volume of 8 ml/kg in patients who would be ventilated with PCV mode. The number of breaths (Dräger Primus) was adjusted to provide an end-tidal carbon dioxide concentration (etCO2) level of 30-35 mmHg. PEEP was set to 5 cmH2O.
  Interventions: Procedure: Pressure controlled ventilation (PCV) mode

INTERVENTIONS:
Procedure: Volume controlled ventilation (VCV) mode — Patients to be ventilated with VCV mode were placed on respiratory support (Dräger Primus) with a breathing rate that would provide 8 ml/kg tidal volume, 5 cmH2O PEEP, and 30-35 mmHg end-tidal carbon dioxide concentration (etCO2) level.
  Lung ultrasonography was performed at 4 different time periods (before laryngeal mask airway (LMA), at the 10th minute after LMA, before extubation and at the 10th minute after extubation). Modified lung ultrasonography scores of 12 quadrants were recorded.
  Arms: Patients ventilated with volume controlled ventilation (VCV) mode
Procedure: Pressure controlled ventilation (PCV) mode — Appropriate peak inspiratory pressure was set to create a tidal volume of 8 ml/kg in patients who would be ventilated with PCV mode. The number of breaths (Dräger Primus) was adjusted to provide an end-tidal carbon dioxide concentration (etCO2) level of 30-35 mmHg. PEEP was set to 5 cmH2O.
  Lung ultrasonography was performed at 4 different time periods (before laryngeal mask airway (LMA), at the 10th minute after LMA, before extubation and at the 10th minute after extubation). Modified lung ultrasonography scores of 12 quadrants were recorded.
  Arms: Patients ventilated with pressure controlled ventilation (PCV) mode

SUMMARY:
General anesthesia is characterized by temporary loss of consciousness and decreased reflex activity without any change in vital functions. It can be performed with intravenous and/or inhalation agents. During general anesthesia, breathing is stopped and respiratory support is provided to patients with various respiratory equipment and ventilation modes on the anesthesia device. The most commonly used ventilation modes during anesthesia are volume controlled (VCV) and pressure controlled (PCV). In pressure-controlled ventilation, ventilation is provided with the airway pressure determined by the anesthesiologist throughout inspiration. While the pressure is constant during inspiration, the tidal volume is variable. In volume controlled ventilation, ventilation executed at the volume is set by the anesthesiologist. In other words, the determined volume is constant, but airway pressures vary.

In pediatric anesthesia practice modes have not been shown to have a clear advantage over each other. Both modes have advantages and disadvantages. With the development of modern anesthesia devices in recent years, safe ventilation can be provided even in very young children with volume controlled mode (VCV).

Atelectasis is the restriction of gas exchange due to complete or partial collapse of the lung. Atelectasis can be seen in 90 percent of patients receiving general anesthesia. This incidence is reported to be 68-100 percent in children.

Lung ultrasonography is an imaging method with many advantages for imaging lung-related diseases, such as not containing ionizing radiation, being inexpensive, and being performed at the bedside. Recently, its use by anesthesiologists has become widespread in many lung pathologies, including atelectasis. Traditional and modified lung ultrasonography scoring systems can be used to evaluate atelectasis in lung parenchyma with ultrasonography. In addition to the traditional system, modified scoring system also enables to evaluate small subpleural consolidations

In this study, it was aimed to compare the effects of volume controlled and pressure controlled ventilation modes used in general anesthesia in children on atelectasis with lung ultrasonography.

DETAILED DESCRIPTION:
Traditional and modified lung ultrasonography scoring systems can be used to evaluate atelectasis in the lung parenchyma by ultrasonography. The modified scoring system also provides the opportunity to evaluate small subpleural consolidations in addition to the traditional system.

Lung tissue is evaluated between the intercostal spaces. On ultrasound, the pleural line can usually be seen as bright white due to the acoustic impedance difference between the aerated lung tissue and the surrounding tissues. Most of the ultrasound waves are reflected from this line. Due to the constantly reflected ultrasound waves between the pleural line and the transducer, hyperechoic lines parallel to the pleural line, called A lines, can be observed in the parenchyma. Vertical hyperechoic lines emerging from the pleural line in the lung ultrasound image are defined as B lines. B lines follow perpendicular to A lines. B lines accompany the sliding movement of the lungs along with the respiratory movement.

The patient is usually evaluated while lying in the supine position. The thorax is divided into 12 quadrants when evaluated with ultrasound for atelectasis. Midsternal line, anterior axillary line, posterior axillary line form the vertical boundaries of the quadrants. Each area is divided into two parts, upper and lower, by a line passing through its midpoint. Left hemithorax anterior upper, lateral upper, posterior upper, anterior lower, lateral lower, posterior lateral; The right hemithorax consists of 12 quadrants: anterior upper, lateral upper, posterior upper, anterior lower, lateral lower, and posterior lateral. The ultrasound probe is advanced transversely and each quadrant is examined. The patient may be asked to turn slightly to the side to evaluate the posterior quadrants. The ultrasound probe is placed vertically on the ribs and the lung parenchyma seen between the intercostal spaces is evaluated. Loss of ventilation is evaluated according to the modified lung ultrasonography scoring system for each quadrant. The score is collected by evaluating 12 quadrants from 0 to 3 and a value between 0-36 is obtained. For each quadrant, 0 represents the region with no ventilation loss and 3 indicates the region with severe ventilation loss. 0 indicates normal tissue with no loss of ventilation and 2 or fewer B lines are observed. 1 indicates little loss of ventilation, 3 or more B lines or one or more subpleural consolidations separated by a normal pleural line are observed. 2 indicates moderate loss of ventilation, observed as multiple fused B lines or multiple small subpleural consolidations separated by thickened or irregular pleural lines. 3 indicates severe loss of ventilation and is observed as consolidation or subpleural consolidation larger than 1x2 cm.

Each patient underwent transthoracic lung ultrasonography a total of 4 times: before laryngeal mask airway (LMA), at the 10th minute after LMA, before extubation and at the 10th minute after extubation. In addition, data on respiratory mechanics and hemodynamic parameters were recorded twice, at the 10th minute after LMA and before extubation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 and 10 years old
* American Society of Anesthesiologists (ASA) Scoring I-II
* Elective surgery planned
* Cases that will undergo general anesthesia
* Surgical time is expected to be >30 minutes

Exclusion Criteria:

* Patients who are allergic to ultrasonography (USG) gel
* Known obstructive and restrictive lung disease
* Pulmonary infection in the last 3 months
* Having a history of surgery in the last 3 months
* A history of multiple trauma in the last 3 months
* Body Mass Index ≥30
* With diaphragmatic hernia
* Having undergone laparoscopic abdominal surgery

Ages: 24 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Volume-controlled ventilation (VCV ) and pressure-controlled ventilation (PCV) respiratory ventilation modes modified lung ultrasonography scores before extubation | Before extubation
  Comparison of the total modified lung ultrasonography score of 12 quadrants (0-36 points) before extubation between groups in terms of atelectasis. An increase in the USG score indicates an increase in the severity of atelectasis. A decrease in the USG score indicates that the severity of atelectasis is low.

SECONDARY OUTCOMES:
Frequency of atelectasis in volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) respiratory ventilation modes | Before LMA (preoperative period)
  Determining the frequency of atelectasis in all quadrants before laryngeal mask airway (LMA) (preoperative period) and comparing it between the two groups
Frequency of atelectasis in volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) respiratory ventilation modes | 10th minute after LMA
  Determining the frequency of atelectasis in all quadrants in the 10th minute after LMA and comparing it between the two groups
Frequency of atelectasis in volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) respiratory ventilation modes | 10th minute after extubation
  Determining the frequency of atelectasis in all quadrants in the 10th minute after extubation and comparing it between the two groups
Comparison of atelectasis incidence and modified Lung ultrasonography (USG) scores (0-3 points) in 12 different lung regions of patients followed in VCV/PCV ventilation modes under general anesthesia. | pre-LMA period (preoperative period), 10th minute after LMA, pre-extubation period, 10th minute after extubation
  The frequency of atelectasis in all lung quadrants in the pre-LMA period, at the 10th minute after LMA, in the pre-extubation period, and at the 10th minute after extubation will be determined and compared.An increase in the USG score indicates an increase in the severity of atelectasis. A decrease in the USG score indicates that the severity of atelectasis is low.
The effects of these ventilation modes on lung pressures parameters. | 10th minute after LMA, pre-extubation period
  Effect of different ventilation modes on lung pressures (peak pressure cmH2O, plat pressure cmH2O, and mean pressure cmH2O parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Aras, MD, Principal Investigator — Republic of Türkiye Ministry of Health Ankara Etlik City Hospital
Locations (1):
- Ahmet Aras, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No